CLINICAL TRIAL: NCT05008198
Title: Assessing an Electroencephalography (EEG) Biomarker of Response to Transcranial Magnetic Stimulation for Major Depression
Brief Title: Assessing an EEG Biomarker of Response to TMS for Major Depression
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Providence VA Medical Center (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); White River Junction Veterans Affairs Medical Center (U.S. Federal Agency); Emory University (Other); University of California, Los Angeles (Other); Edward Hines Jr. VA Hospital (U.S. Federal Agency); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); VA Pittsburgh Healthcare System (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CSDR-001-19S
Record Dates: First submitted 2021-07-30; First posted 2021-08-17 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: depression; transcranial magnetic stimulation; electroencephalography; biomarkers
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transcranial Magnetic Stimulation: Transcranial Magnetic Stimulation is delivered as part of routine care and is not managed by this observational study.
  Interventions: Other: Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation is delivered as part of routine care and is not managed by this observational study.
  Other Names: TMS; Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Veterans with treatment resistant depression (TRD) have the opportunity to receive transcranial magnetic stimulation (TMS) treatment via the VA's National TMS Clinical Pilot Program. While some see improvement with their depression, others do not. Therefore, it may be beneficial to be able to predict with biomarkers what participants may see improvement with their treatment. Electroencephalography (EEG) is a means to identify such biomarkers. Four hundred Veterans with TRD will be enrolled in this trial to determine whether neuroimaging biomarkers of repetitive transcranial magnetic stimulation (TMS) can be prospectively replicated in a large ecologically valid sample. Participants will have a total of EEG scans at baseline, every 5th treatment session, and at the end of treatment for a total of 7 EEG scans.

DETAILED DESCRIPTION:
The goals of this study are to: (1) test a potential predictive resting EEG biomarker of antidepressant response (differential patters of gamma oscillations) in a large sample of Veterans with TRD receiving TMS (N=400); (2) assess whether a second putative biomarker (early changes in theta cordance during treatment) predict eventual response to TMS, as well as, leverage this large sample to identify other potential biomarkers (such as markers of early versus late response to TMS, markers of response to other TMS parameters (e.g., 5 Hz, 1 Hz or theta burst TMS), and markers of change with treatment that may speak to mechanism); and (3) create an infrastructure to rapidly identify and test additional EEG-based biomarkers of treatment response in patients with depression and other psychiatric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Veterans participating in the VA TMS Pilot Program age 18 years or older
* Able to provide written informed consent to participate in the EEG portion of this study and to allow linking such data to data collected as part of the TMS Pilot Program
* Diagnosis of MDD based on DSM-5 criteria and be currently depressed despite prior treatment with at least one adequate antidepressant treatment
* Receiving stable doses of psychiatric medications (no dose changes for >4 weeks prior to study entry), in stable psychotherapy, or receiving no psychiatric medications and/or psychotherapy

Exclusion Criteria:

* History of seizure disorder
* Known structural or neurologic abnormalities present or close to the treatment site that would increase risk of seizure
* History of brain surgery
* History of recent traumatic brain injury (within 6 months) or any history of moderate to severe traumatic brain injury
* Clinical evidence of severe or uncontrolled alcohol or substance use disorders within three months
* Active withdrawal from alcohol or other substances of abuse
* Implanted metal device in the head that would increase the risk of TMS
* Metal in the head that would increase the risk of TMS
* Current psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with major depressive disorder (MDD) participating in the VA Clinical TMS Pilot Program. Given the complex nature of the Veteran population, the primary diagnosis of MDD may be comorbid with other disorders, including post-traumatic stress disorder (PTSD).
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Inventory of Depressive Symptomatology-Self Report (IDS-SR) | 1) Baseline, pre-treatment and 2) 6 weeks, treatment completion
  The IDS-SR is a 30-item self-report depressive symptom severity rating scale. The IDS-SR has been shown to have highly acceptable psychometric properties and has been found to be a treatment sensitive measures of symptom severity in depression. Each question is on a scale of 0 to 4. The IDS-SR has a score range between 0 to 84, with a higher score reflecting higher symptom severity in depression.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Holtzheimer, MD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (1):
- White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT05008198/ICF_000.pdf